CLINICAL TRIAL: NCT03227224
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, Adaptive Dose-Finding Study to Evaluate the Efficacy and Safety of JNJ-42847922 as Adjunctive Therapy to Antidepressants in Adult Subjects With Major Depressive Disorder Who Have Responded Inadequately to Antidepressant Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of JNJ-42847922 as Adjunctive Therapy to Antidepressants in Adult Participants With Major Depressive Disorder Who Have Responded Inadequately to Antidepressant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108281; 42847922MDD2001 (Other: Janssen Research & Development, LLC); 2015-005282-22 (EudraCT Number)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive 2 placebo capsules matching JNJ-42847922 once daily orally from Day 1 to Day 41 (Week 6).
  Interventions: Drug: Placebo
- JNJ-42847922 (Experimental): Participants will receive 2 capsules of JNJ-42847922 once daily orally from Day 1 to Day 41 (Week 6).
  Interventions: Drug: JNJ-42847922

INTERVENTIONS:
Drug: Placebo — Participants will receive 2 placebo capsules matching JNJ-42847922 once daily orally from Day 1 to Day 41 (Week 6).
  Arms: Placebo
Drug: JNJ-42847922 — Participants will receive 2 capsules of JNJ-42847922 once daily orally from Day 1 to Day 41 (Week 6).
  Other Names: MIN-202;; Seltorexant
  Arms: JNJ-42847922

SUMMARY:
The purpose of this study is to assess the dose-response relationship of 2 doses of JNJ-42847922 before interim analysis, and potentially 3 doses based on interim analysis results, compared to placebo as adjunctive therapy to an antidepressant drug in improving depressive symptoms in participants with Major Depressive Disorder (MDD) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI); and to assess the safety and tolerability of JNJ-42847922 compared to placebo as adjunctive therapy to an antidepressant in participants with MDD.

DETAILED DESCRIPTION:
The study will investigate the antidepressant effects of a range of doses of JNJ-42847922 (seltorexant) (versus placebo), as adjunctive treatment to antidepressant drugs for treatment of MDD, and will assess the safety and tolerability of JNJ-42847922. The study will be conducted in 3 phases: a screening phase (up to 4 weeks), a double-blind treatment phase (6 weeks), and a post-treatment follow-up phase (2 weeks). Efficacy, safety, pharmacokinetic, and biomarker evaluations will be performed in the study at defined timepoints. The duration of the study will be up to approximately 12 weeks (84 days).

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential (WONCBP), aged 18 to 70 years (inclusive). A WONCBP is defined as: a).Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. b). Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy. c). If reproductive status is questionable, additional evaluation should be considered
* Meet Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Structured Clinical Interview for DSM-5 Axis I Disorders- Clinical Trials Version (SCID-CT). In addition their major depressive episode must be deemed "valid" using the SCID Screening Questionnaire (SSQ) interview administered by remote, independent raters. The length of the current depressive episode must be less than or equal to (<=) 18 months
* Have had an inadequate response to at least 1 but no more than 3 antidepressants, administered at an adequate dose and duration in the current episode of depression, as measured by the Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ). An inadequate response is defined as less than (<)50 percent (%) reduction in depressive symptom severity, as assessed by the MGH-ATRQ. An adequate trial is defined as an antidepressant treatment for at least 4 weeks at or above the minimum therapeutic dose specified in the MGH-ATRQ, for any particular antidepressant. The inadequate response must include the participant's current antidepressant treatment
* Participants receiving monotherapy treatment for depressive symptoms with one of the following selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants, in any formulation: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at or above the minimum therapeutic dose level) for at least 4 weeks, and for no greater than 12 months, at screening. Modification of an effective preexisting therapy should not be made for the explicit purpose of entering a subject into the study
* Have a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=)25 (performed by independent, centralized remote raters) at screening and must not demonstrate a clinically significant improvement (that is, an improvement of greater than [>]20% on their MADRS total score) from the screening to baseline visit
* Must be otherwise healthy on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening. If the results of the clinical laboratory tests are outside the normal reference ranges, the participant could be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Has a history of, or current signs and symptoms of, severe renal insufficiency (creatinine clearance <30 milliliter per minute [mL/min]); moderate to severe hepatic insufficiency (Child-Pugh Score 7-9), significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic (including narcolepsy), hematologic, rheumatologic, immunologic or endocrine disorders (including uncontrolled hypo- or hyperthyroidism or diabetes, or insulin-dependent diabetes mellitus). Participants with non-insulin dependent diabetes mellitus who are well-controlled (hemoglobin A1C [HbA1C] <=7.5% and fasting glucose <126 milligram per deciliter [mg/dL] at screening) could be eligible to participate if otherwise medically healthy, and if on a stable regimen of glucose-lowering medications for at least 2 months prior to screening
* Has signs and symptoms of Cushing's Disease, Addison's Disease, primary amenorrhea, or other evidence of significant medical disorders of the hypothalamic-pituitary-adrenal (HPA) axis
* Has a history of lack of response to 3 or more adequate antidepressant treatments, as indicated by no or minimal (<= 25% improvement in symptoms) when treated with an antidepressant of adequate dose (per MGH-ATRQ) and duration (at least 4 weeks)
* Has history or current diagnosis of a psychotic disorder, bipolar disorder, mental retardation, autism spectrum disorder, or borderline personality disorder, somatoform disorders, chronic fatigue syndrome or fibromyalgia
* Has any significant primary sleep disorder, including but not limited to obstructive sleep apnea, restless leg syndrome, or parasomnias

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (101):
- United States (33):
  - California Pharmaceutical Research Institute, Inc., Anaheim, California
  - Catalina Research Institute, Chino, California
  - Synergy Clinical Research Center Of Escondido, Lemon Grove, California
  - Asclepes Research, Panorama City, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - SF-Care, Inc, San Rafael, California
  - Collaborative NeuroScience Network, Torrance, California
  - Elite Clinical Trials, Wildomar, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Clinical NeuroScience Solutions Inc, Jacksonville, Florida
  - Innovative Clinical Research Inc, Lauderhill, Florida
  - Qps-Mra, Llc, Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - Behavioral Clinical Research , Inc, North Miami, Florida
  - Clinical NeuroScience Solutions Inc, Orlando, Florida
  - Compass Research LLC, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Radiant Research, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Clinilabs, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Clinical Trials of America, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Neuro Behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Core Clinical Research, Everett, Washington
- Bulgaria (14):
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - State Psychiatric Hospital Kardzhali, Kardzhali
  - State Psychiatric Hospital - Lovech, Lovech
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - MC 'Hipokrat - N', EOOD, Plovdiv
  - Mental Health Center - Rousse, Rousse
  - MHC - Sofia, EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment - UMHAT Alexandrovska EAD, Sofia
  - Medical Center 'Doverie', Sofia
  - Medical Center Intermedica, OOD, Sofia
  - MHAT-Targovishte, AD, Targovishte
  - State Psychiatric Hospital - Tzarev Brod, Tzarev Brod
  - Diagnostic Consulting Center Mladost - M Varna, Varna
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
- Finland (4):
  - Mederon Oy, Helsinki
  - Savon Psykiatripalvelu, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu, Rauma
- France (5):
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Cabinet Medical des Drs Prizac-Desbonnet Scottez, Douai
  - CHU Nimes Hopital Caremeau, Nîmes
  - Hopital Sainte Anne, Paris
  - Centre Hospitalier Guillaume Regnier, Rennes
- Germany (4):
  - Neurologische Praxis Dr. Schoell & Kollegen, Bad Homburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Somni Bene GmbH, Schwerin
- Japan (18):
  - Hongo Todaimae Mental Clinic, Bunkyō City
  - Kuramitsu Hospital, Fukuoka
  - National Center for Global Health and Medicine Kohnodai hospital, Ichikawa-shi
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki-gun
  - Nara Medical University Hospital, Kashihara-shi
  - Senzoku Mental Clinic, Meguro-ku
  - Heart Care Ginga Clinic, Nakano
  - Shiranui Hospital, Omuta-shi
  - Seiwakai Yutaka Clinic, Sagamihara-shi
  - Sangenjaya Nakamura Mental Clinic, Setagaya-ku
  - Yoyogi Mental Clinic, Shibuya-ku
  - Etoh Mental Clinic, Shinagawa-ku
  - Nishi-Shinjuku Concieria Clinic, Shinjuku-ku
  - Tamaki Clinic, Shinjuku-ku
  - Shinjuku Research Park Clinic, Shinjuku-ku
  - Ohwa Mental Clinic, Toshima-ku
  - Sekino Hospital, Toshima-ku
  - Jisenkai Hozumi Himorogi Clinic, Toshima-ku
- Russia (13):
  - SHI Arkhangelsk Regional Clinical Psychiatric Hospital, Arkhangelsk
  - City Clinical Psychiatric Hopsital 3, Moscow
  - FSI Moscow SRI of Psychiatry of Minzdravsocrazvitia, Moscow
  - Closed corporation 'Scientific Center of Personalized Psychiatry', Moscow
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow
  - Clinical Psychiatry Hospital n.a. N.N. Solodovnikov, Omsk
  - Medical and Rehabilitation Research Center Phoenix, Rostov-on-Don
  - City Psychiatric Hospital of St. Nikolay Chudotvorets, Saint Petersburg
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Engels psychiatric hospital, Saratov Region
  - Research Institute of Mental Health, Tomsk
  - Sverdlov Regional Psychiatric Clinical Hospital, Yekaterinburg
- Ukraine (10):
  - CNCE'Precarpathian Regional Clinical Mental Health Center Ivano-Frankivsk RC', Ivano-Frankivsk
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - Cnce 'Kyiv City Psychoneurological Hospital #2' of Executive Body of Kyiv City Council (Kcsa), Kyiv
  - CNCE of the Lviv Regional Council 'Lviv Regional Clinical Psychiatric Hospital', Lviv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - CNCE Odesa regional psychiatric hospital #2 Odesa regional council, Oleksandrivka
  - Poltava O.F. Maltsev RC Psychiatric Hospital Dept #9 (Ad-P Dept) HSEIU Ukrainian MSA, Poltava
  - Ternopil RCCPH Depts of Psychiatry #2 (m) & Psychiatry #4 (f) Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - CI O.I. Yuschenko VRPsH Depts #7 & #10 M.I. Pyrogov VNMU, Vinnytsia
  - CNCE 'Vinnytsya RC Psychoneurological Hospital n.a. O.I. Yushchenko Vinnytsya RC', Vinnytsia

REFERENCES:
- [Derived] Savitz A, Wajs E, Zhang Y, Xu H, Etropolski M, Thase ME, Drevets WC. Efficacy and Safety of Seltorexant as Adjunctive Therapy in Major Depressive Disorder: A Phase 2b, Randomized, Placebo-Controlled, Adaptive Dose-Finding Study. Int J Neuropsychopharmacol. 2021 Dec 8;24(12):965-976. doi: 10.1093/ijnp/pyab050. PMID 34324636

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants in the double-blind treatment period received seltorexant matching placebo capsule once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Seltorexant 10 mg: Participants in the double-blind treatment period received seltorexant 10 milligrams (mg) capsules once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Seltorexant 20 mg: Participants in the double-blind treatment period received seltorexant 20 mg capsules once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Seltorexant 40 mg: Participants in the double-blind treatment period received seltorexant 40 mg capsules (2*20 mg capsules) once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
Period: Double-blind Treatment Period (6 Weeks)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Started | 138 | 33 | 63 | 53
Treated | 137 | 33 | 61 | 52
Completed | 123 | 27 | 55 | 46
Not Completed | 15 | 6 | 8 | 7
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Received a Disallowed Concomitant Treatment | 0 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 4
Not completed — Non-Compliance with Study Drug | 2 | 1 | 0 | 1
Not completed — Other | 4 | 0 | 1 | 0
Period: Follow-up Phase (2 Weeks)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Started | 138 (All participants that started the double-blind period were followed-up for follow-up phase.) | 33 (All participants that started the double-blind period were followed-up for follow-up phase.) | 63 (All participants that started the double-blind period were followed-up for follow-up phase.) | 53 (All participants that started the double-blind period were followed-up for follow-up phase.)
Completed | 134 | 29 | 57 | 50
Not Completed | 4 | 4 | 6 | 3
Not completed — Other | 4 | 4 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg | Total
Number analyzed (Participants) | 137 | 33 | 61 | 52 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.71) | 49.4 (15.31) | 48.5 (13.56) | 48.3 (10.52) | 49.1 (12.34)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 131 | 29 | 59 | 51 | 270
  From 65 to 84 years | 6 | 4 | 2 | 1 | 13
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 20 | 30 | 28 | 152
  Male | 63 | 13 | 31 | 24 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 3 | 9 | 8 | 40
  Black or African American | 11 | 1 | 2 | 5 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White | 105 | 29 | 50 | 39 | 223
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 1 | 5 | 7 | 28
  Not Hispanic or Latino | 120 | 31 | 53 | 42 | 246
  Unknown or Not Reported | 2 | 1 | 3 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  BULGARIA | 35 | 2 | 17 | 12 | 66
  FINLAND | 3 | 1 | 1 | 5 | 10
  GERMANY | 0 | 1 | 1 | 1 | 3
  JAPAN | 18 | 3 | 8 | 8 | 37
  RUSSIAN FEDERATION | 18 | 16 | 8 | 3 | 45
  UKRAINE | 22 | 6 | 6 | 5 | 39
  UNITED STATES | 41 | 4 | 20 | 18 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition.
Time Frame: Baseline to Week 6
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 124 | 26 | 55 | 47
score on a scale | -12.3 (10.95) | -12.2 (8.33) | -15.0 (12.13) | -14.7 (13.29)
Statistical Analysis 1: Comparison: Placebo vs Seltorexant 10 mg; Test type: Superiority; p = 0.724, Mixed model for repeated measures (MMRM); Difference of Least Square Means = 0.9, 90% CI 2-sided [-3.12 to 4.82]
Statistical Analysis 2: Comparison: Placebo vs Seltorexant 20 mg; Test type: Superiority; p = 0.083, MMRM; Difference of Least Square Means = -3.1, 90% CI 2-sided [-6.13 to -0.16]
Statistical Analysis 3: Comparison: Placebo vs Seltorexant 40 mg; Test type: Superiority; p = 0.424, MMRM; Difference of Least Square Means = -1.5, 90% CI 2-sided [-4.70 to 1.63]

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between the initial administration of study drug and 2 days after the last administration of study drug.
Time Frame: Up to Week 8
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 137 | 33 | 61 | 52
percentage of participants | 40.9 | 33.3 | 41.0 | 36.5

3. Primary Outcome: Percentage of Participants With Clinically Significant Laboratory Abnormalities
Description: Percentage of participants with clinically significant laboratory abnormalities were reported which included Gamma-glutamyl transferase (GGT), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), Creatine Kinase (CK), Lactate Dehydrogenase (LDH), Albumin , bicarbonate, bilirubin, calcium, chloride, cholesterol, creatinine, direct bilirubin, glucose, high density lipoprotein (HDL) cholesterol, hemoglobin A1C, low density lipoprotein (LDL) cholesterol, phosphate, potassium, protein, sodium, triglycerides, urate, and urea nitrogen.
Time Frame: Up to Week 8
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; n (number analyzed) signifies those participants who were evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 137 | 31 | 61 | 52
percentage of participants
  ALT: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  ALT: Abnormally high | 0 | 0 | 0 | 1.9
  Albumin: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 52
  Albumin: Abnormally low | 0 | 0 | 0 | 0
  Albumin: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Albumin: Abnormally high | 0 | 0 | 0 | 0
  ALP: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  ALP: Abnormally high | 0 | 0 | 0 | 0
  AST: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 51
  AST: Abnormally high | 0 | 0 | 0 | 0
  Bicarbonate: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 52
  Bicarbonate: Abnormally low | 0 | 0 | 0 | 0
  Bicarbonate: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Bicarbonate: Abnormally high | 0 | 0 | 0 | 0
  Bilirubin: Abnormally high | 0 | 0 | 0 | 0
  Calcium: Abnormally low | 0 | 0 | 0 | 0
  Calcium: Abnormally high | 0 | 0 | 0 | 0
  Chloride: Abnormally low: number analyzed (Participants) | 134 | 31 | 60 | 52
  Chloride: Abnormally low | 0.7 | 0 | 0 | 0
  Chloride: Abnormally high: number analyzed (Participants) | 134 | 31 | 60 | 52
  Chloride: Abnormally high | 0 | 0 | 0 | 0
  Cholesterol: Abnormally high: number analyzed (Participants) | 131 | 29 | 56 | 51
  Cholesterol: Abnormally high | 0 | 0 | 0 | 0
  CK: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  CK: Abnormally high | 0 | 0 | 1.7 | 0
  Creatinine: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Creatinine: Abnormally high | 0 | 0 | 0 | 0
  Direct Bilirubin: Abnormally high: number analyzed (Participants) | 134 | 31 | 60 | 51
  Direct Bilirubin: Abnormally high | 0 | 0 | 0 | 0
  GGT: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  GGT: Abnormally high | 0 | 0 | 0 | 0
  Glucose: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 51
  Glucose: Abnormally low | 0 | 0 | 0 | 0
  Glucose: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 51
  Glucose: Abnormally high | 0 | 0 | 0 | 0
  HDL Cholesterol: Abnormally low: number analyzed (Participants) | 131 | 29 | 55 | 51
  HDL Cholesterol: Abnormally low | 2.3 | 6.9 | 1.8 | 2.0
  Hemoglobin A1C: Abnormally low: number analyzed (Participants) | 132 | 28 | 57 | 51
  Hemoglobin A1C: Abnormally low | 0.0 | 0 | 0 | 0
  Hemoglobin A1C: Abnormally high: number analyzed (Participants) | 132 | 28 | 57 | 51
  Hemoglobin A1C: Abnormally high | 0 | 0 | 0 | 0
  LDL Cholesterol: Abnormally low: number analyzed (Participants) | 131 | 29 | 54 | 51
  LDL Cholesterol: Abnormally low | 4.6 | 10.3 | 9.3 | 5.9
  LDL Cholesterol: Abnormally high: number analyzed (Participants) | 131 | 29 | 54 | 51
  LDL Cholesterol: Abnormally high | 7.6 | 6.9 | 1.9 | 11.8
  LDH: Abnormally high: number analyzed (Participants) | 133 | 31 | 60 | 51
  LDH: Abnormally high | 0 | 0 | 0 | 0
  Phosphate: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 51
  Phosphate: Abnormally low | 0.7 | 3.2 | 3.3 | 7.8
  Phosphate: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 51
  Phosphate: Abnormally high | 0 | 0 | 0 | 0
  Potassium: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 51
  Potassium: Abnormally low | 0 | 0 | 0 | 0
  Potassium: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 51
  Potassium: Abnormally high | 0.7 | 3.2 | 0 | 0
  Protein:Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 52
  Protein:Abnormally low | 0 | 0 | 0 | 0
  Sodium: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 52
  Sodium: Abnormally low | 0 | 0 | 0 | 0
  Sodium: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Sodium: Abnormally high | 0 | 0 | 0 | 0
  Triglycerides: Abnormally high: number analyzed (Participants) | 131 | 29 | 55 | 51
  Triglycerides: Abnormally high | 0 | 0 | 0 | 0
  Urate: Abnormally low: number analyzed (Participants) | 135 | 31 | 60 | 52
  Urate: Abnormally low | 0 | 0 | 0 | 0
  Urate: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Urate: Abnormally high | 0 | 0 | 5.0 | 1.9
  Urea Nitrogen: Abnormally high: number analyzed (Participants) | 135 | 31 | 60 | 52
  Urea Nitrogen: Abnormally high | 0 | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Vital Signs (Systolic Blood Pressure [SBP] and Diastolic Blood Pressure [DBP]) at Day 8
Description: Change from baseline in vital signs (SBP and DBP) at Day 8 was reported.
Time Frame: Baseline and Day 8
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
millimeters of mercury (mmHg)
  Standing DBP | -0.7 (6.29) | -0.5 (5.22) | 0.7 (5.86) | 0.9 (6.41)
  Standing SBP | -0.4 (8.16) | -0.8 (7.19) | 0.2 (8.17) | 0.3 (9.71)
  Supine DBP | -0.8 (6.32) | -0.9 (6.19) | 2.3 (6.14) | 1.2 (6.67)
  Supine SBP | 0.1 (8.19) | 1.6 (6.56) | 1.5 (9.57) | 0.5 (10.19)

5. Primary Outcome: Change From Baseline in Vital Signs (SBP and DBP) at Day 22
Description: Change from baseline in vital signs (SBP and DBP) at Day 22 was reported.
Time Frame: Baseline and Day 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 132 | 29 | 58 | 49
mmHg
  Standing DBP | 0.0 (6.67) | -1.2 (5.92) | -0.4 (6.90) | 2.4 (7.42)
  Standing SBP | 0.2 (7.01) | -1.2 (6.55) | -2.7 (9.62) | 1.6 (11.29)
  Supine DBP | -0.4 (6.81) | -1.8 (6.7) | -0.2 (7.41) | 2.6 (6.81)
  Supine SBP | 0.8 (8.14) | 0.3 (4.76) | -0.9 (10.78) | 2.2 (10.08)

6. Primary Outcome: Change From Baseline in Vital Signs (SBP and DBP) at Day 42
Description: Change from baseline in vital signs (SBP and DBP) at Day 42 was reported.
Time Frame: Baseline and Day 42
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 126 | 28 | 56 | 48
mmHg
  Standing DBP | -0.5 (6.22) | 0.3 (9.16) | -0.8 (6.75) | 2.9 (7.96)
  Standing SBP | -0.5 (7.99) | 1.1 (7.92) | -3.2 (10.57) | 2.0 (9.9)
  Supine DBP | -0.6 (7.1) | -1.6 (9.23) | 0.0 (8.31) | 2.1 (7.5)
  Supine SBP | 0.6 (8.88) | -0.5 (10.00) | -1.3 (10.85) | 1.9 (8.35)

7. Primary Outcome: Change From Baseline in Vital Signs (SBP and DBP) at Endpoint (Week 6)
Description: Change from baseline in vital signs (SBP and DBP) at endpoint was reported.
Time Frame: Baseline and Endpoint (Week 6)
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure. Endpoint (double-blind [DB]) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
mmHg
  Standing DBP | -0.3 (6.29) | 0.6 (8.98) | -0.6 (6.78) | 2.8 (7.79)
  Standing SBP | -0.3 (8.33) | 1.0 (7.42) | -3.1 (10.29) | 1.8 (9.89)
  Supine DBP | -0.4 (7.08) | -1.4 (9.34) | 0.2 (8.35) | 2.3 (7.39)
  Supine SBP | 0.6 (8.81) | -0.3 (9.38) | -1.4 (10.52) | 1.6 (8.58)

8. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate [PR]) at Day 8
Description: Change from baseline in vital sign (PR) at Day 8 was reported.
Time Frame: Baseline and Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
Beats per minute
  Standing PR | -0.1 (7.95) | -0.7 (7.07) | 0.9 (9.17) | 1.3 (9.21)
  Supine PR | 0 (7.15) | -1.2 (7.16) | 0.5 (6.23) | 1.7 (9.32)

9. Primary Outcome: Change From Baseline in Vital Sign (PR) at Day 22
Description: Change from baseline in vital sign (PR) at Day 22 was reported.
Time Frame: Baseline and Day 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 132 | 29 | 58 | 49
Beats per minute
  Standing PR | 1.4 (7.57) | 0.7 (7.36) | 1.5 (8.27) | 0.3 (9.59)
  Supine PR | 1.5 (7.61) | -0.7 (7.31) | 2.8 (7.94) | 0.9 (10.55)

10. Primary Outcome: Change From Baseline in Vital Sign (PR) at Day 42
Description: Change from baseline in vital sign (PR) at Day 42 was reported.
Time Frame: Baseline and Day 42
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 126 | 28 | 56 | 48
Beats per minute
  Standing PR | 0.8 (7.99) | -1.4 (9.35) | 1.5 (8.99) | -0.6 (9.04)
  Supine PR | 0.3 (8.16) | -2.8 (8.67) | 2.4 (9.01) | -0.6 (9.71)

11. Primary Outcome: Change From Baseline in Vital Sign (PR) at Endpoint (Week 6)
Description: Change from baseline in vital sign (PR) at endpoint (Week 6) was reported.
Time Frame: Baseline and Endpoint (Week 6)
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
Beats per minute
  Standing PR | 0.4 (8.4) | -1.6 (9.27) | 2.1 (9.34) | -0.5 (9.11)
  Supine PR | 0.2 (8.16) | -2.4 (8.97) | 2.4 (8.78) | -0.5 (9.60)

12. Primary Outcome: Change From Baseline in Vital Sign (Temperature) at Day 8
Description: Change from baseline in vital Sign (temperature) at Day 8 was reported.
Time Frame: Baseline and Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
Celsius | -0.01 (0.324) | -0.05 (0.274) | 0.02 (0.278) | 0.06 (0.300)

13. Primary Outcome: Change From Baseline in Vital Sign (Temperature) at Day 22
Description: Change from baseline in vital Sign (temperature) at Day 22 was reported.
Time Frame: Baseline and Day 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 132 | 29 | 58 | 48
Celsius | -0.02 (0.299) | -0.01 (0.242) | -0.02 (0.332) | 0.02 (0.392)

14. Primary Outcome: Change From Baseline in Vital Sign (Temperature) at Day 42
Description: Change from baseline in vital Sign (temperature) at Day 42 was reported.
Time Frame: Baseline and Day 42
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 126 | 28 | 56 | 48
Celsius | 0.02 (0.326) | -0.04 (0.291) | -0.05 (0.223) | 0.05 (0.445)

15. Primary Outcome: Change From Baseline in Vital Sign (Temperature) at Endpoint (Week 6)
Description: Change from baseline in vital Sign (temperature) at endpoint (Week 6) was reported.
Time Frame: Baseline and Endpoint (Week 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 52
Celsius | 0.02 (0.317) | -0.03 (0.276) | -0.06 (0.242) | 0.06 (0.437)

16. Primary Outcome: Change From Baseline in Physical Examination (Waist Circumference) at Day 42
Description: Change from baseline in physical examination (waist circumference) was reported.
Time Frame: Baseline and Day 42
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 32 | 58 | 51
centimeters (cm) | 0.31 (2.778) | -0.50 (1.972) | 0.00 (3.523) | -0.48 (9.498)

17. Primary Outcome: Change From Baseline in Physical Examination (Body Weight) at Day 42
Description: Change from baseline in physical examination (body weight) was reported.
Time Frame: Baseline and Day 42
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 32 | 58 | 51
Kilograms (kg) | 0.19 (2.373) | 0.01 (1.889) | 0.05 (1.563) | 0.61 (1.946)

18. Primary Outcome: Change From Baseline in Physical Examination (Body Mass Index [BMI]) at Day 42
Description: Change from baseline in physical examination (BMI) was reported.
Time Frame: Baseline and Day 42
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 32 | 58 | 51
kilograms per meter square (kg/m^2) | 0.07 (0.850) | 0.01 (0.662) | 0.02 (0.553) | 0.22 (0.715)

19. Primary Outcome: Percentage of Participants With Treatment-emergent Abnormal Electrocardiogram (ECG) Values Outside Pre-defined Limits
Description: Percentage of participants with treatment-emergent abnormal ECG values (Heart rate less than or equal to [<=] 50 or greater than or equal to [>=] 100 beats per minute [bpm], PR interval <=120 or >=200 milliseconds [msec], QRS interval <=60 or >=120 msec, and QT interval <=200 or >=500 msec) outside pre-defined limits were reported.
Time Frame: Up to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 30 | 58 | 50
percentage of participants
  Heart rate (<=50) | 0.7 | 0 | 3.4 | 6.0
  Heart rate (>=100) | 0.7 | 0 | 1.7 | 0
  PR interval (<=120) | 0.7 | 0 | 0 | 0
  PR interval (>=200) | 0.7 | 0 | 1.7 | 6.0
  QRS interval (<=60) | 0 | 0 | 0 | 0
  QRS interval (>=120) | 0 | 3.3 | 0 | 0
  QT interval (<=200): number analyzed (Participants) | 134 | 30 | 58 | 49
  QT interval (<=200) | 0 | 0 | 0 | 0
  QT interval (>=500): number analyzed (Participants) | 134 | 30 | 58 | 49
  QT interval (>=500) | 0 | 3.3 | 0 | 0

20. Primary Outcome: Percentage of Participants With Most Severe Post-baseline Potentially Suicide-Related Category Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a clinician-rated instrument that reports severity of both suicidal ideation and behavior. Suicidal ideation was classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. Minimum total score 0, maximum total score 5; higher total scores indicate more suicidal ideation and/or suicidal behavior. If no events qualify for score of 1 to 10, score of 0 was assigned (0= "no event that can be assessed on the basis of C-SSRS"). Higher scores indicate greater severity.
Time Frame: Up to Week 8
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
percentage of participants
  No Event | 94.9 | 96.9 | 96.7 | 94.1
  Suicidal ideation | 5.1 | 3.1 | 3.3 | 5.9
  Suicidal behavior | 0 | 0 | 0 | 0

21. Primary Outcome: Change From Baseline in Sexual Functioning as Measured by Arizona Sexual Experiences Scale (ASEX) Score at Day 42
Description: Effect on sexual functioning was assessed using the ASEX score. The ASEX is a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Each of the 5 items is rated on a 6-point scale, ranging from 1 to 6. The 5 items are summed to create a total score, ranging from 5 to 30, with the higher scores indicating more sexual dysfunction.
Time Frame: Baseline and Day 42
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 133 | 31 | 58 | 49
score on a scale | -1.4 (4.55) | -2.2 (3.62) | -2.4 (4.55) | -2.5 (4.94)

22. Primary Outcome: Physician Withdrawal Checklist-20 (PWC-20) Total Score at Day 43
Description: Intensity of discontinuation symptoms was assessed (for example: underlying depression; anxiety-nervousness; dysphoric mood/depression; difficulty concentrating; weakness; fatigue-lethargy-lack of energy; irritability), using the Physician Withdrawal Checklist (PWC-20) administered by a trained clinician/rater. Symptoms are rated on a scale 0 (No symptom present) and 3 (severe symptoms). Total scores range from 0 to 24 calculated by adding the scores of following 8 items: Nausea-Vomiting, Diarrhea, Poor Coordination, Diaphoresis, Tremor-Tremulousness, Dizziness-Lightheadedness, Increased Acuity Sound Smell Touch, Paresthesias. Higher scores indicating more severe symptoms.
Time Frame: Day 43
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 29 | 58 | 49
score on a scale | 0.9 (1.68) | 0.2 (0.6) | 0.7 (1.6) | 0.5 (0.87)

23. Secondary Outcome: Change From Baseline in the MADRS Total Score by Baseline Insomnia Severity Index (ISI) Score at Day 42
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. The ISI has 7 questions, each rated on a 5-point Likert scale ranging from 0 to 4. The total score is calculated as the sum of the 7 items ranging from 0 to 28. Higher scores represent a more severe condition.
Time Frame: Baseline and Day 42
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specific category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 124 | 26 | 55 | 47
score on a scale
  Day 42: Baseline ISI score per IWRS less than (<)15: number analyzed (Participants) | 50 | 21 | 23 | 13
  Day 42: Baseline ISI score per IWRS less than (<)15 | -13.3 (10.83) | -12.6 (8.01) | -13.0 (11.38) | -14.9 (12.14)
  Day 42: Baseline ISI score per IWRS>=15: number analyzed (Participants) | 74 | 5 | 32 | 34
  Day 42: Baseline ISI score per IWRS>=15 | -11.6 (11.06) | -10.4 (10.41) | -16.5 (12.62) | -14.6 (13.87)

24. Secondary Outcome: Change From Baseline in ISI Total Score at DB Endpoint (Up to Week 6)
Description: The ISI is a commonly used, 7-item psychometrically validated measure used to rate insomnia. Each item is scored 0 (no problem) to 4 (very big problem) with total between 0-28 which is calculated by adding the scores of all 7 items (absence of insomnia [0-7]; sub-threshold insomnia [8-14]; moderate insomnia [15-21]; and severe insomnia [22-28]). The change in ISI total score from baseline at DB endpoint was evaluated. Negative change in score indicates improvement.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies the evaluable participants for this outcome measure. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 134 | 31 | 58 | 51
Units on a scale | -6.3 (6.73) | -4.9 (6.22) | -8.7 (6.91) | -8.5 (8.73)

25. Secondary Outcome: Percentage of Participants With Response on Depressive Symptoms Scale Based on MADRS Total Score
Description: Responders are defined as participants with a >=50 percent (%) improvement in the MADRS total score from baseline to a given timepoint. MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. Participants with missing values at a given time point were imputed as non-responders.
Time Frame: Day 42
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 137 | 33 | 61 | 52
Percentage of participants | 28.5 | 24.2 | 41.0 | 38.5

26. Secondary Outcome: Percentage of Participants With Remission of Depressive Symptoms Based on MADRS Total Score
Description: Participants with a MADRS total score of less than or equal to (<=) 8, <=10, and <=12 at a given time point were considered as remitters. MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. Participants with missing values at a given time point were imputed as non-responders.
Time Frame: Day 42
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 137 | 33 | 61 | 52
Percentage of participants
  MADRS (<=12) | 19.0 | 15.2 | 29.5 | 26.9
  MADRS (<=10) | 17.5 | 9.1 | 26.2 | 26.9
  MADRS (<=8) | 16.1 | 6.1 | 23.0 | 19.2

27. Secondary Outcome: Change From Baseline in Structured Interview Guide for the Hamilton Anxiety Rating Scale (HAM-A) Total Score at Day 42
Description: HAM-A is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. Each of the 14-items in the scale is scored on a 5-point scale, ranging from 0 (a complete lack of that symptom) to 4 (a very severe show of anxiety with that symptom). The total score ranges from 0 to 56 which is calculated by adding the scores of all 14 items, where 0-13 indicates normal range, 14-17 indicates mild severity, 18 -24: mild to moderate severity, 25 -30: moderate to severe, and >=31: severe. Higher score indicates worsening. Negative change in score indicates improvement.
Time Frame: Baseline and Day 42
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies the evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 126 | 27 | 56 | 47
Units on a scale | -8.7 (7.92) | -9.9 (5.57) | -9.6 (9.31) | -9.9 (10.17)

28. Secondary Outcome: Percentage of Participants With Response on Anxiety Symptoms Scale Based on HAM-A Total Score
Description: Participants with a >=50 percent improvement in the HAM-A total score from baseline at a given timepoint were considered as responders. HAM-A is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. Each of the 14-items in the scale is scored on a 5-point scale, ranging from 0 (a complete lack of that symptom) to 4 (a very severe show of anxiety with that symptom). The total score ranges from 0 to 56 which is calculated by adding the scores of all 14 items, where 0-13 indicates normal range, 14-17 indicates mild severity, 18 -24: mild to moderate severity, 25 -30: moderate to severe, and >=31: severe. Higher score indicates worsening. Participants with missing values at a given time point were imputed as non-responders.
Time Frame: Day 42
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 137 | 33 | 61 | 52
Percentage of participants | 37.2 | 57.6 | 50.8 | 46.2

29. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at DB Endpoint (Up to Week 6)
Description: The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of illness exhibited by a participant, rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores indicate worsening. Negative change in score indicates improvement.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 135 | 30 | 60 | 52
Units on a scale | -1.0 [-5 to 2] | -1.0 [-3 to 1] | -1.0 [-5 to 1] | -1.0 [-5 to 1]

30. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Score at Day 42
Description: The SDS is a 5-item questionnaire which has been widely used and accepted for assessment of functional impairment and associated disability. The first 3 items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0-10 rating scale. The scores for the first 3 items are summed to create a total score of 0-30, where a higher score indicates greater impairment. It also has 1 item on days lost from school or work and 1 item on days when underproductive. Negative change in score indicates improvement.
Time Frame: Baseline and Day 42
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 96 | 16 | 30 | 26
Units on a scale | -7.9 (6.99) | -7.5 (5.19) | -7.9 (7.46) | -5.9 (9.20)

31. Secondary Outcome: Change From Baseline in the MADRS Total Score at Day 42 in Participants With Major Depressive Disorder (MDD) With Anxious Distress Versus Participants With MDD Without Anxious Distress
Description: MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score range of 0-60 which is calculated by adding the scores of all 10 items. Higher scores represent a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline and Day 42
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (numbers of participants analyzed) signifies numbers of participants evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specific category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 124 | 26 | 55 | 46
Units on a scale
  MDD with Anxious Distress: number analyzed (Participants) | 76 | 13 | 31 | 31
  MDD with Anxious Distress | -13.9 (11.50) | -11.0 (8.67) | -16.9 (12.31) | -15.3 (13.0)
  MDD without Anxious distress: number analyzed (Participants) | 48 | 13 | 24 | 15
  MDD without Anxious distress | -9.7 (9.59) | -13.4 (8.15) | -12.5 (11.70) | -13.8 (14.63)

32. Secondary Outcome: Change From Baseline in Salivary Cortisol Levels, Measured Upon Awakening at Days 8, 22 and 42
Description: Exposure on the hypothalamic-pituitary-adrenal (HPA) axis in participants with MDD was evaluated by assessing change in salivary cortisol levels.
Time Frame: Baseline, Days 8, 22 and 42
Population: Biomarker analysis set included all randomized participants who received at least 1 dose of study drug during the double-blind phase and had biomarker data at baseline. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specific timepoints.
Measure: Mean (Standard Deviation); unit: nanomoles per Liter (nmol/L)
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 117 | 26 | 48 | 38
nanomoles per Liter (nmol/L)
  Change at Day 8: number analyzed (Participants) | 116 | 26 | 48 | 38
  Change at Day 8 | 0.2 (8.41) | 0.7 (7.24) | 0.0 (8.64) | -0.4 (6.19)
  Change at Day 22: number analyzed (Participants) | 117 | 21 | 45 | 38
  Change at Day 22 | 0.4 (8.65) | 2.1 (6.39) | 0.7 (6.75) | 1.0 (10.75)
  Change at Day 42: number analyzed (Participants) | 112 | 18 | 45 | 37
  Change at Day 42 | 1.0 (10.85) | 1.5 (6.15) | -1.2 (6.67) | -0.5 (6.69)

33. Secondary Outcome: Plasma Concentrations of Seltorexant and Its Metabolites (M12 and M16)
Description: Plasma concentrations of Seltorexant and its metabolites (M12 and M16) over time were reported.
Time Frame: Day 1: Between 0.25 hours (h) to 1.5 hour, 2 to 4 hours, and 6 to 8 hours post-dose; Day 8 (morning): 6 to 12 hours post evening dose of Day 7
Population: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specific timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 28 | 59 | 50
nanograms per milliliter (ng/mL)
  Seltorexant: Day 1, 0.25h-1.5h: number analyzed (Participants) | 24 | 46 | 43
  Seltorexant: Day 1, 0.25h-1.5h | 181 (165) | 277 (291) | 535 (500)
  Seltorexant: Day 1, 2-4h: number analyzed (Participants) | 24 | 46 | 43
  Seltorexant: Day 1, 2-4h | 199 (113) | 374 (232) | 647 (325)
  Seltorexant: Day 1, 6-8h: number analyzed (Participants) | 24 | 46 | 43
  Seltorexant: Day 1, 6-8h | 117 (99.3) | 167 (179) | 207 (169)
  Seltorexant: Day 8, Morning (6 to 12 hours post evening dose of Day 7) | 52.8 (65.8) | 69.4 (119) | 104 (203)
  M12: Day 1,0.25h-1.5h: number analyzed (Participants) | 24 | 46 | 43
  M12: Day 1,0.25h-1.5h | 118 (107) | 194 (223) | 357 (367)
  M12: Day 1, 2-4h: number analyzed (Participants) | 24 | 46 | 43
  M12: Day 1, 2-4h | 146 (58.8) | 283 (185) | 513 (284)
  M12: Day 1, 6-8h: number analyzed (Participants) | 24 | 46 | 43
  M12: Day 1, 6-8h | 105 (73.5) | 187 (189) | 279 (278)
  M12: Day 8, Morning (6 to 12 hours post evening dose of Day 7) | 76.2 (79) | 99 (133) | 169 (251)
  M16: Day 1, 0.25h-1.5h: number analyzed (Participants) | 24 | 46 | 43
  M16: Day 1, 0.25h-1.5h | 29.1 (30.2) | 47 (53.4) | 71.4 (78.3)
  M16: Day 1, 2-4h: number analyzed (Participants) | 24 | 46 | 43
  M16: Day 1, 2-4h | 33.3 (15.7) | 61.4 (35.7) | 101 (49.3)
  M16: Day 1, 6-8h: number analyzed (Participants) | 24 | 46 | 43
  M16: Day 1, 6-8h | 27.5 (16.6) | 40.1 (31.4) | 70.6 (33.6)
  M16: Day 8, Morning (6 to 12 hours post evening dose of Day 7) | 23.7 (14.9) | 37.6 (36.1) | 61.7 (43.7)

34. Secondary Outcome: Change From Baseline in Depressive Symptoms Using the Patient Health Questionnaire 9-Item (PHQ-9) at DB Endpoint (Up to Week 6)
Description: The PHQ-9 is a 9-item, Patient Reported Outcome (PRO) measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participants item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19) and Severe (20-27).
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | -7.3 (6.14) | -6.2 (5.48) | -8.6 (6.66) | -7.0 (7.64)

35. Secondary Outcome: Change From Baseline in Anhedonia Using the Snaith-Hamilton Pleasure Scale (SHAPS) Score at DB Endpoint (Up to Week 6)
Description: The SHAPS is a 14-item, self-report instrument to assess hedonic capacity in adults with MDD. Each of the items has a set of 4 response categories-Definitely Agree (=1), Agree (=2), Disagree (=3), and Definitely Disagree (=4). A total score is created with either of the Disagree responses receiving a score of 1 and either of the Agree responses receiving a score of 0. The participants item responses are summed to provide a total score ranging from 0 to 14. A higher total SHAPS score indicates higher levels of current anhedonia.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | -3.6 (4.44) | -2.3 (4.09) | -4.2 (4.50) | -3.2 (5.20)

36. Secondary Outcome: Change From Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form at DB Endpoint (Up to Week 6)
Description: The PROMIS-SD Short Form subscale consists of a static 8 item questionnaire. It assesses the concepts of sleep initiation (2 items), quality of sleep (3 items), early morning feelings (2 items) and worrying about sleep (1 item). Responses to each of the 8 items range from 1 to 5, and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS-SD indicate more of the concept measured (disturbed sleep). Negative change in score indicates improvement.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | -6.4 (8.53) | -5.1 (8.39) | -10.2 (9.21) | -10.9 (9.25)

37. Secondary Outcome: Change From Baseline in Fatigue Using the Patient Reported Outcome Measurement Information System-Fatigue (PROMIS-F) Short Form Subscale Score at DB Endpoint (Up to Week 6)
Description: The PROMIS-Fatigue Short Form subscale consists of a static 8 item questionnaire. It assesses a range of symptoms from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Ratings are done on a 5-item Likert scale ranging from 0 (not at all) to 5 (very much) or 0 (never) to 5(always) depending upon the question answered. Higher scores on the PROMIS-F indicate more of the concept measured (fatigue). Negative change in score indicates improvement.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | -7.7 (8.45) | -7.4 (8.25) | -9.4 (8.62) | -8.0 (10.29)

38. Secondary Outcome: Change From Baseline in Severity of Depression Using the Patient Global Impression-Severity (PGI-S) Score at DB Endpoint (Up to Week 6)
Description: The PGI-S is a self-report scale to measure severity of illness (1=none, 2=mild, 3=moderate, 4=severe). Higher score indicates more illness severity. Negative change in score indicates improvement.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: as for outcome 35
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | -1.0 [-3 to 2] | 0.0 [-2 to 1] | -1.0 [-3 to 1] | -1.0 [-3 to 1]

39. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) Heath State Index Total Score at DB Endpoint (Up to Week 6)
Description: EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D-5L dimensions were scored using a utility-weighted algorithm to derive an EQ-5D-5L health status index score between 0 (death) to 100 (full health).
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | 0.188 (0.2201) | 0.143 (0.1856) | 0.229 (0.2084) | 0.158 (0.2841)

40. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analog Scale (VAS) Total Score at Endpoint (Up to Week 6)
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It consists of the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ-VAS). EQ-5D-5L (describing and valuing health-related quality of life) descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the participant's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. Higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement. EQ-VAS self-rating records respondent's own assessment of his/her overall health status at time of completion, on scale of 0 (worst health you can imagine) to 100 (best health you can imagine).
Time Frame: Baseline and Endpoint (up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Endpoint (DB) values: last measurement within double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 136 | 32 | 60 | 51
Units on a scale | 17.4 (20.55) | 8.9 (19.34) | 23.4 (21.18) | 20.1 (23.08)

41. Secondary Outcome: Change From Baseline in Work Productivity and Limitations Using the Work Limitations Questionnaire (WLQ) Short Form Score at DB Endpoint (Up to Week 6)
Description: The WLQ is to assess the on-the-job impact of chronic health problems and/or treatment ("work limitations") in adults. It is a 8-item questionnaire self-report rating scale developed to measure the on-the-job impact of chronic health problems and/or treatment ("work limitations"). It comprises five dimensions of limitations: handling time, physical, mental-interpersonal, productivity loss and output demands. Participants respond to each item with options ranging from 'Almost all of the time' to 'none of the time', or 'Does not apply to my job'. Each dimension of limitations have a scale score ranging from 0 to 100 with lower score indicating low level of work limitations.
Time Frame: Baseline and DB Endpoint (Up to Week 6)
Population: Full analysis set included participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure; 'n' (number analyzed) signifies those participants who were evaluable for specific categories. Endpoint (DB) values are from the last measurement within the double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 109 | 31 | 34 | 34
Units on a scale
  Time management: number analyzed (Participants) | 104 | 31 | 22 | 32
  Time management | -21.3 (30.41) | -18.2 (28.28) | -21.8 (34.46) | -20.8 (37.48)
  Physical demands: number analyzed (Participants) | 105 | 25 | 33 | 34
  Physical demands | -15.2 (23.64) | -23.5 (26.10) | -11.7 (31.4) | -14.3 (35.37)
  Mental interpersonal scale: number analyzed (Participants) | 109 | 25 | 34 | 33
  Mental interpersonal scale | -21.2 (27.61) | -19.5 (25.28) | -26.28 (27.89) | -15.9 (31.76)
  Output demand scale: number analyzed (Participants) | 103 | 22 | 32 | 30
  Output demand scale | -23.9 (26.72) | -22.2 (27.8) | -20.3 (30.08) | -21.7 (35.80)
  Productivity loss: number analyzed (Participants) | 99 | 31 | 29 | 29
  Productivity loss | -5.1 (5.56) | -4.7 (5.30) | -4.7 (6.16) | -4.6 (7.02)

42. Primary Outcome: Physician Withdrawal Checklist-20 (PWC-20) Total Score From Day 49 to Day 56
Description: as for outcome 22
Time Frame: Day 49 to Day 56
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Seltorexant 10 mg | Seltorexant 20 mg | Seltorexant 40 mg
Number analyzed (Participants) | 133 | 29 | 57 | 50
score on a scale | 0.9 (1.91) | 0.4 (0.78) | 0.8 (1.64) | 0.7 (1.25)

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: Safety analyses set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug.
Groups:
- Double-blind: Seltorexant 10 mg: Participants in the double-blind treatment period received Seltorexant 10 milligrams (mg) capsules once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Double-blind: Seltorexant 20 mg; Follow-up: Seltorexant 20 mg: Participants in the double-blind treatment period received seltorexant 20 mg capsules once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- DB: Seltorexant 40 mg; Follow-up: Seltorexant 40 mg: Participants in the double-blind treatment period received seltorexant 40 mg capsules (2*20 mg capsules) once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Follow-up: Placebo: Participants in the double-blind treatment period received matching placebo capsule once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
- Follow-up: Seltorexant 10 mg: Participants in the double-blind treatment period received seltorexant 10 mg capsules once daily orally from Day 1 to Day 41 (Week 6). Participants had a follow-up visit within 7 to 14 days after double-blind treatment period. During the follow-up phase, participants were followed-up for the safety assessments on Day 43 (Week 7).
Arm/Group | Placebo | Double-blind: Seltorexant 10 mg | Double-blind: Seltorexant 20 mg | DB: Seltorexant 40 mg | Follow-up: Placebo | Follow-up: Seltorexant 10 mg | Follow-up: Seltorexant 20 mg | Follow-up: Seltorexant 40 mg
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/33 | 0/61 | 0/52 | 0/137 | 0/33 | 0/61 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/137 | 0/33 | 0/61 | 0/52 | 0/137 | 0/33 | 0/61 | 0/52
Other Adverse Events (participants affected / at risk) | 22/137 | 5/33 | 11/61 | 12/52 | 1/137 | 0/33 | 0/61 | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | Double-blind: Seltorexant 10 mg (N=33) | Double-blind: Seltorexant 20 mg (N=61) | DB: Seltorexant 40 mg (N=52) | Follow-up: Placebo (N=137) | Follow-up: Seltorexant 10 mg (N=33) | Follow-up: Seltorexant 20 mg (N=61) | Follow-up: Seltorexant 40 mg (N=52)
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=137) | Double-blind: Seltorexant 10 mg (N=33) | Double-blind: Seltorexant 20 mg (N=61) | DB: Seltorexant 40 mg (N=52) | Follow-up: Placebo (N=137) | Follow-up: Seltorexant 10 mg (N=33) | Follow-up: Seltorexant 20 mg (N=61) | Follow-up: Seltorexant 40 mg (N=52)
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 4 | 3 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 2 | 1 | 6 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 7 | 1 | 6 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03227224/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03227224/SAP_001.pdf